CLINICAL TRIAL: NCT04618107
Title: Principal Investigator
Brief Title: Wide Awake Surgery for Tendon Repair in Hand Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Saba Kiran, Principal investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1316
Record Dates: First submitted 2020-10-31; First posted 2020-11-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-10

CONDITIONS: Tendon Injury - Hand
MeSH Terms: interventions — Anesthesia, General

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wide awake surgery (Experimental): Wide awake local anaesthesia was used as mode of aneasthesia for tendon repair surgery. Functional outcome of in terms of active range of motion was calculated via Strickland method and American Society for the surgery of the hand criteria at sixth week of surgery using goniometer
  Interventions: Procedure: Wide awake surgery
- General anaesthesia (Active Comparator): Tendon repair surgeries were performed under general anaesthesia. Functional outcome of in terms of active range of motion was calculated via Strickland method and American Society for the surgery of the hand criteria at sixth week of surgery using goniometer
  Interventions: Procedure: General anaesthesia

INTERVENTIONS:
Procedure: Wide awake surgery — Wide awake local anaesthesia was used to perform tendon repair surgeries.Local anaesthetic injections given using 27 gauze needle in subcutaneous tissue plane.Tendon repair performed using modified Kessler repair.Outcome of surgery assesed at sixth postoprative week.
  Arms: Wide awake surgery
Procedure: General anaesthesia — Tendon repair performed under general anaesthesia using modified Kessler repair.Outcomes of surgery assesed at sixth post operative week
  Arms: General anaesthesia

SUMMARY:
Wide awake surgery for tendon repair in hand trauma To compare the functional outecomes in terms of active range of motion for tendon repair surgeries performed under wide awake anaesthesia versus general anaesthesia.

DETAILED DESCRIPTION:
All patients aged 15 or above with hand trauma resulting in tendon injuries were included.65 patients undergoing tendon repair in wide awake anaesthesia were grouped as approach arm and another 65 patients of general anaesthesia group were kept as control arm.Range of motion of corresponding tendons were measured at completion of sixth postoperative week using goniometer.Total active range of motion were calculated according to criteria given by Strickland method and American Society for Surgery ofthe Hand (ASSH).

Functional outcomes were compared among two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of either gender of age 15 years or above.
2. All of the patients with hand injuries with tendon repair required, operated within the hospital premises

Exclusion Criteria:

1. Patients allergic to agents of local anesthesia.
2. Patients with anxiety symptoms
3. Patients with mental disorders rendering them unable to comprehend and follow intraoperative commands.
4. Patients with associated nerve injuries.
5. Patients requiring bone fixation or with other complex injuries and with soft tissue loss requiring coverage.
6. Patients with massive contamination, crush injuries or infection which needs to be addressed and treated prior to definitive repair.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
active range of motion | six weeks
  active range of motion assesd by strickland and American Society for surgery criteria

CONTACTS AND LOCATIONS:
Overall Officials: Saba Kiran, MBBS, Principal Investigator — Dow University of Health Sciences
Locations (1):
- Saba Kiran, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Neill N, Abdall-Razak A, Norton E, Kumar A, Shah H, Khatkar H, Alsafi Z, Agha R. Use of Wide-Awake Local Anaesthetic No Tourniquet (WALANT) in upper limb and hand surgery: A systematic review protocol. Int J Surg Protoc. 2020 Mar 13;20:8-12. doi: 10.1016/j.isjp.2020.03.001. eCollection 2020. PMID 32258835
- [Background] Fulchignoni C, Bonetti MA, Rovere G, Ziranu A, Maccauro G, Pataia E. Wide awake surgery for flexor tendon primary repair: A literature review. Orthop Rev (Pavia). 2020 Jun 25;12(Suppl 1):8668. doi: 10.4081/or.2020.8668. eCollection 2020 Jun 29. PMID 32913601
- [Background] Libberecht K, Lafaire C, Van Hee R. Evaluation and functional assessment of flexor tendon repair in the hand. Acta Chir Belg. 2006 Sep-Oct;106(5):560-5. doi: 10.1080/00015458.2006.11679952. PMID 17168270